CLINICAL TRIAL: NCT03556449
Title: High Resolution Ultrasound of Scapulae Alatae - Correlation With Electrophysiological Measurements - a Prospective Case Control Study
Brief Title: High Resolution Ultrasound of Scapulae Alatae - a Prospective Case Control Study
Status: Completed | Type: Observational
Sponsor: Sándor Beniczky (Other)
Responsible Party: Sponsor-Investigator, Sándor Beniczky, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: USSA; 3532 (Other Grant/Funding Number: The Lundbeck Foundation); 1-10-72-152-18 (Other: The regional Committee on Health Research Ethics, Denmark)
Record Dates: First submitted 2018-05-24; First posted 2018-06-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2018-06

CONDITIONS: Scapula Alata; Scapular Winging
Keywords: scapula/innervation*; Thoracic Nerves/injuries*; Peripheral Nerve Injuries; Shoulder; Musculoskeletal Diseases/diagnosis*
MeSH Terms: conditions — Wounds and Injuries; Peripheral Nerve Injuries; Musculoskeletal Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: High resolution ultrasound
  Interventions: Diagnostic Test: High resolution ultrasound
- Healthy subjects: High resolution ultrasound
  Interventions: Diagnostic Test: High resolution ultrasound

INTERVENTIONS:
Diagnostic Test: High resolution ultrasound — Using a high-frequency linear array transducer (18L6 HD)
  Other Names: Siemens ACUSON S1000

SUMMARY:
Scapula alata, caused by disturbance in the scapulothoracic stabilizer muscles due to nerve injury, is a relatively rare but also underreported disease. It can lead to years of invalidity of the affected upper extremity, considerable pain and social and emotional consequences for the patients. Unrecognized and misdiagnosed scapula alata and, consequently, wrong or delayed treatment is a general problem in this patient group. Today the diagnosis is based on the clinical examination and the electrophysiological examination. One of the problems is that the electrophysiological examination in a fair part of the patients is not showing any pathology even though the history of the patient and the clinical evaluation are indicating scapula alata.

This study is a single-blinded, prospective, controlled multicentre study. The aim of the study is to investigate whether ultrasound can be used as a supplement to the electrophysiological examination when diagnosing scapula alata. Ultrasound will be used to visualize possible thickening of the cross-sectional area of nerves and the degree and pattern of muscle involvement in patients with scapula alata. By comparing measurements from scapula alata patients with the measurements from healthy controls, we are able to see if ultrasound can distinguish these two groups from each other. Furthermore, we will examine whether the ultrasound measurements correlate with the electrophysiological findings in patients and, when available, compare the ultrasound measurements of muscle thickness with MRI (magnetic resonance Imaging) findings. The use of ultrasound in scapula alata patients may help determine the presence and severity of a nerve lesion and the subsequent degree of muscle involvement and may therefore serve as a supplement to the clinical diagnosis.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Clinical suspicion of scapula alata

Exclusion Criteria:

* Winged scapula due to other cause than nerve damage. eg. myopathy

Healthy subjects

Exclusion Criteria:

* History of Shoulder trauma or shoulder disease
* History of cervical radiculopathy
* History of upper extremity peripheral neuropathy/plexopathy
* Peripheral vascular disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients: From patients referred to the department of Neurophysiology, Aarhus University hopsital.
  Healthy subjects: From recruitment posters at Aarhus University, Aarhus University Hospital and at http://www.forsoegsperson.dk/.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Thickness of musculus serratus anterior | 10-15 minuttes
Thickness of musculus trapezius | 10-15 minuttes
Thickness of musculus rhomboideus | 10-15 minuttes
Cross sectional area of nervus thoracicus longus | 10-15 minuttes
Cross sectional area of nervus accesorius | 10-15 minuttes
Cross sectional area of nervus dorsalis scapularis | 10-15 minuttes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Neurophysiology, the department of Neurology, Aarhus University Hospital, Aarhus, Denmark